CLINICAL TRIAL: NCT00002561
Title: A Phase III Study of Radiotherapy or ABVD Plus Radiotherapy Versus ABVD Alone in the Treatment of Early Stage Hodgkin's Disease
Brief Title: Radiation Therapy and Chemotherapy in Treating Patients With Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HD6; CAN-NCIC-HD6 (Other: PDQ); E-JHD06 (Other: ECOG); NCI-V94-0427 (Other Grant/Funding Number: NCI); CDR0000063481 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-11-21 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hodgkin Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Bleomycin; Dacarbazine; Doxorubicin; Vinblastine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy or ABVD + Radiotherapy (Active Comparator): Radiotherapy
  Interventions: Biological: bleomycin sulfate; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine; Radiation: radiation therapy
- ABVD Alone (Active Comparator): ABVD Alone
  Interventions: Biological: bleomycin sulfate; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine

INTERVENTIONS:
Biological: bleomycin sulfate — 10 units/m2
Drug: dacarbazine — 375mg/m2
Drug: doxorubicin hydrochloride — 25mg/m2
Drug: vinblastine — 6mg/m2
Radiation: radiation therapy — 35Gy in 20 fractions (daily)
  Arms: Radiotherapy or ABVD + Radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high energy x-rays to damage tumor cells. Combining more than one drug or combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy, with or without chemotherapy, with chemotherapy alone in treating patients with stage I or stage IIA Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the 12-year survival of patients with clinical stage I-IIA Hodgkin's disease treated with radiotherapy with or without doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) versus ABVD only. II. Compare the freedom from progression at 5 and 10 years in patients treated with these regimens. III. Compare the complete remission rate, freedom from secondary disease progression at 5 and 10 years, and cause-specific survival at 5, 10, and 15 years in patients treated with these regimens. IV. Compare the short- and long-term toxicity of these regimens in these patients. V. Compare the quality of life of patients in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center. Patients who are under age 40 and have lymphocyte-predominant or nodular sclerosing histology, an erythrocyte sedimentation rate less than 50, and fewer than 4 disease sites (supradiaphragmatic or pelvic node sites) are assigned to cohort 1 (good prognosis). All other patients are assigned to cohort 2 (poor prognosis). Cohort 1: Arm I: Patients with supradiaphragmatic disease undergo radiotherapy to the supradiaphragmatic lymph node areas (mantle region), spleen, and para-aortic lymph nodes 5 days a week for 4 weeks. Patients with pelvic disease undergo radiotherapy to an "inverted-Y" field (excluding the spleen) 5 days a week for 4 weeks. Arm II: Patients receive doxorubicin, bleomycin, vinblastine, and dacarbazine IV on days 1 and 15 (ABVD). Treatment continues every 4 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Patients with complete remission (CR) after course 2 receive 2 additional courses past CR. Patients with partial remission (PR) after course 2 receive 4 additional courses past PR. Patients with unconfirmed/uncertain complete remission (CRu) receive 2-4 additional courses past CRu. Cohort 2: Arm III: Patients receive ABVD as in arm II, followed 4-6 weeks later by concurrent radiotherapy to the mantle region and upper abdomen to the level of L2 5 days a week for 4 weeks. Alternatively, radiotherapy may also be administered sequentially to the mantle region 5 days a week for 4 weeks and then to the upper abdomen to the level of L2 5 days a week for 4 weeks. Arm IV: Patients receive ABVD only as in arm II. Patients with disease progression after treatment in arms II or IV are considered for radiotherapy. Quality of life is assessed on day 1 of each course of chemotherapy (arms II-IV) and on day 28 of the last course of chemotherapy (arms II and IV); on the first and final days of radiotherapy (arms I and III); at 4 weeks and at 3, 6, and 12 months after completion of radiotherapy (arms I and III) or chemotherapy (arms II and IV); and then annually for 2-10 years. Patients are followed at months 3, 6, and 12 and then annually thereafter.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study within 7.5 years.

ELIGIBILITY:
Eligibility Criteria

* Histologically proven Hodgkin's Disease. A needle aspirate specimen will not be considered sufficient for diagnosis.
* Pathologic material must have been reviewed by a designated local reference pathologist (LRP) prior to randomization. Histologic subtype determined by the LRP will be used for patient cohort assignment.
* Patients must have clinical stage I - IIA disease according to Ann Arbor staging criteria. Clinical stage must be based on at least one tissue biopsy. The following aspects are to be considered in determining patient stage:

  i) Splenic Enlargement: Splenic enlargement determined by imaging studies only should not be considered evidence of splenic involvement with Hodgkin's disease. Patients should be considered as having splenic involvement if the spleen is palpable on physical examination and enlarged on imaging studies, or imaging studies show focal abnormalities consistent with Hodgkin's disease. These patients, if presenting with supradiaphragmatic disease would therefore be assessed as having Stage III disease and would be ineligible.

ii) Bone Disease: Lytic or blastic lesions seen on plain radiographs or abnormalities on bone scan consistent with Hodgkin's disease will be considered as bone involvement with Hodgkin's disease. These patients would therefore be assessed as having Stage IV disease and would be ineligible.

iii) Pleural Effusion and Ascites: The presence of a pleural effusion or ascites will be considered as evidence of Hodgkin's disease even if cytological examination is negative. These patients would be assessed as having probable Stage IV disease and therefore would be ineligible. Patients assessed on Xray as having pleural thickening or "blunting" of the costophrenic angle only may be eligible. iv) Extra-nodal vs. Stage IV Disease: Patients with disease involving a single extra-nodal site may be considered as "limited-stage" provided all disease can be included in a standard radiation field. Patients with extra-nodal disease that cannot be included in such a field (eg, lung, bone) or with multiple sites of extra-nodal disease are not eligible for this trial.

* Pulmonary function tests must be done in patients with symptomatic lung disease. FVC, FEV-1 and DLCO must be ≥ 60% of predicted value. Patients with asthma controlled by medication are eligible if the above criteria are met.
* Patient's age is ≥ 16 years. (Note that the lower age limit at each centre will be determined by that centre's policy regarding the age at which an individual may sign their own consent.)
* Patient must not have received previous chemotherapy or radiotherapy.
* Laboratory requirements:

granulocytes ≥ 1.5 x 109/L (S.I.) or ≥ 1.5 x 103/uL (U.S.) platelets ≥ 125 x 109/L (S.I.) or ≥ 125 x 103/uL (U.S.) bilirubin ≤ 2.5 x UNL (unless due to hemolytic anemia) serum creatinine ≤ 2 x UNL

* Patient must have been seen by both a radiation oncologist and medical oncologist who agree the patient is able to receive protocol radiation therapy.
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Clinical Trials Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is given. The patient must sign the consent form prior to randomization. Please note that the consent form for this study must contain a statement which gives permission for the NCICCTG and monitoring agencies to review patient records.
* Availability of patient for follow-up and quality of life (QoL) assessments. Patients must be accessible for treatment and follow-up. Investigators must assure themselves that patients registered on this trial will be available for complete documentation of the treatment, toxicity and follow-up. Comparison of quality of life is an end-point of this study. Patients must have completed the pre-randomization quality of life assessment and be willing to complete future assessments. The only exceptions will be patients who are unable to read english or french. Patients on study are expected to complete all the quality of life assessments but, should this not prove possible, they will be retained in the study for all other analyses.

Ineligibility Criteria

* Prior or concurrent malignancies, except adequately treated basal cell carcinoma of the skin. (Patients with prior carcinoma-in-situ of the cervix are not eligible.)
* Cardiac disease defined as symptomatic congestive heart failure or coronary artery disease, known valvular (other than asymptomatic mitral valve prolapse) or congenital heart disease (other than asymptomatic atrial septal defects) or need for cardiac medications. Hypertension controlled with drug therapy is not an exclusion criterion.
* Other major medical illness judged likely by the local investigator to preclude safe administration of protocol treatment or required follow-up.
* Patients with stage IA disease (who might be treated with involved-field only irradiation) defined by meeting all of the following criteria:

  i) lymphocyte predominant or nodular sclerosing histology ii) disease bulk < 3 cm iii) erythrocyte sedimentation rate (ESR) < 50 iv) unilateral high - neck only disease, defined as disease located above the upper border of the thyroid cartilage or isolated epitrochlear adenopathy
* Patients with very unfavourable clinical stage I-IIA disease defined as bulky adenopathy. Bulky adenopathy is defined as a palpable nodal mass greater than 10 cm. in diameter or a mediastinal mass with a maximum mass diameter measuring greater than or equal to 1/3 the maximum chest wall diameter (see Appendix III).
* Patients with intra-abdominal disease. (Patients with pelvic disease: ileofemoral, inguinal or parailiac nodes are eligible for this study.)
* Patients with B symptoms.
* Patients known to have a positive antibody test for the human immunodeficiency virus (HIV) or who have a clinical diagnosis of acquired immunodeficiency syndrome. HIV testing is not a requirement for study entry.
* Patients who have undergone a staging laparotomy.
* Female patients who are pregnant. Note: men and women of childbearing age must be advised in the use of adequate contraception.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 1994-01-25 (Actual); Primary Completion 2011-08-15 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Survival | 12 years
  12 year survival comparison

SECONDARY OUTCOMES:
Freedom from progression | 12 years
Complete response rate | 12 years
Second disease progression rate | 5 and 10 years
Cause-specific survival rate | 5 and 10 years
  treatment-related toxicity and Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph M. Meyer, MD, FRCPC, Study Chair — Margaret and Charles Juravinski Cancer Centre; Jane N. Winter, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (22):
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Italy (2):
  - Instituto del Radio O. Alberti Spedali Civili, Brescia
  - Policlinico Monteluce/Univ. Degli Studi Di Perugia, Perugia
- Royal South Hants Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Macdonald DA, Ding K, Gospodarowicz MK, Wells WA, Pearcey RG, Connors JM, Winter JN, Horning SJ, Djurfeldt MS, Shepherd LE, Meyer RM. Patterns of disease progression and outcomes in a randomized trial testing ABVD alone for patients with limited-stage Hodgkin lymphoma. Ann Oncol. 2007 Oct;18(10):1680-4. doi: 10.1093/annonc/mdm287. Epub 2007 Sep 10. PMID 17846017
- [Result] Macdonald DA, Gospodarowicz MK, Wells WA, et al.: Relapse patterns and subsequent outcomes of patients treated on the NCIC CTG HD.6 (ECOG JHD06) randomized trial evaluating ABVD alone in patients with limited stage Hodgkin's lymphoma (HL). [Abstract] Blood 106 (11): A-817, 2005.
- [Result] Meyer RM, Gospodarowicz MK, Connors JM, Pearcey RG, Bezjak A, Wells WA, Burns BF, Winter JN, Horning SJ, Dar AR, Djurfeldt MS, Ding K, Shepherd LE; National Cancer Institute of Canada Clinical Trials Group; Eastern Cooperative Oncology Group. Randomized comparison of ABVD chemotherapy with a strategy that includes radiation therapy in patients with limited-stage Hodgkin's lymphoma: National Cancer Institute of Canada Clinical Trials Group and the Eastern Cooperative Oncology Group. J Clin Oncol. 2005 Jul 20;23(21):4634-42. doi: 10.1200/JCO.2005.09.085. Epub 2005 Apr 18. PMID 15837968
- [Result] Meyer R, Gospodarowicz M, Connors J, et al.: A randomized phase III comparison of single - modality ABVD with a strategy that includes radiation therapy in patients with early-stage Hodgkin's disease: the HD-6 trial of the National Cancer Institute of Canada Clinical Trials Group (Eastern Cooperative Oncology Group Trial JHD06). [Abstract] Blood 102 (11 Pt 1): A-81, 2003.
- [Derived] Hay AE, Klimm B, Chen BE, Goergen H, Shepherd LE, Fuchs M, Gospodarowicz MK, Borchmann P, Connors JM, Markova J, Crump M, Lohri A, Winter JN, Dorken B, Pearcey RG, Diehl V, Horning SJ, Eich HT, Engert A, Meyer RM; Conducted by the NCIC Clinical Trials Group (Canada) and German Hodgkin Study Group (GHSG). An individual patient-data comparison of combined modality therapy and ABVD alone for patients with limited-stage Hodgkin lymphoma. Ann Oncol. 2013 Dec;24(12):3065-9. doi: 10.1093/annonc/mdt389. Epub 2013 Oct 11. PMID 24121121
- [Derived] Meyer RM, Gospodarowicz MK, Connors JM, Pearcey RG, Wells WA, Winter JN, Horning SJ, Dar AR, Shustik C, Stewart DA, Crump M, Djurfeldt MS, Chen BE, Shepherd LE; NCIC Clinical Trials Group; Eastern Cooperative Oncology Group. ABVD alone versus radiation-based therapy in limited-stage Hodgkin's lymphoma. N Engl J Med. 2012 Feb 2;366(5):399-408. doi: 10.1056/NEJMoa1111961. Epub 2011 Dec 11. PMID 22149921